CLINICAL TRIAL: NCT00946504
Title: A Two-Way Crossover Bioequivalence Study Comparing Single 10 mg Doses of Geneva's 10 mg Glipizide Tablets To Roerig's 10 mg Glucotrol Tablets
Brief Title: To Demonstrate the Relative Bioequivalency Comparing Geneva's 10 mg Glipizide Tablets To Roerig's 10 mg Glucotrol Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9208525-G2
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glipizide

ARMS (2):
- 1 (Experimental): Glipizide 10 mg Tablets (Geneva Pharmaceutical, Inc.)
  Interventions: Drug: Glipizide 10 mg Tablets (Geneva Pharmaceutical, Inc.)
- 2 (Active Comparator): Glucotrol 10 mg Tablets (Roerig Pharmaceutical, Inc.)
  Interventions: Drug: Glucotrol 10 mg Tablets (Roerig Pharmaceutical, Inc.)

INTERVENTIONS:
Drug: Glipizide 10 mg Tablets (Geneva Pharmaceutical, Inc.)
  Arms: 1
Drug: Glucotrol 10 mg Tablets (Roerig Pharmaceutical, Inc.)
  Arms: 2

SUMMARY:
To demonstrate the relative bioequivalency comparing Geneva's 10 mg Glipizide tablets to Roerig's 10 mg Glucotrol tablets.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 1992-10; Primary Completion 1992-10 (Actual); Study Completion 1992-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Roger D. Anderson, M.D., Principal Investigator — Biodecision, Inc.